CLINICAL TRIAL: NCT01530165
Title: A Translation Randodomized Trial of Culturally Specific and Cost Effective Life Style Intervention for the Prevention of Type 2 Diabetes in Pakistan
Brief Title: (Pakistan Diabetes Prevention Program PDPP)
Acronym: PDPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: International Diabetes Federation (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Dr. Asma Ahmed, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DS10-A5
Record Dates: First submitted 2011-11-21; First posted 2012-02-09 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Prediabetic State & High Risk Individuals on the Basis of Diabetes Risk Score
Keywords: IFG; IGTT
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Intervention versus Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Pre diabetics randomized to control arm will receive standard life style advice which is given to all pre diabetics seeking medical advice. Group counselling (30 min to 1 hour) will be provided to participants enrolled in control arm in which they will attend one group class at baseline where they will be given basic information on diabetes prevention , weight loss, diet, and exercise consitent with expert recommendations for a healthy life style inclusing losing 5-10% of their excess body weight to reduce their calorie and fat intake and exercising at least 150 minutes per week.
- life style intervention arm (Other): This arm would be given aggressive life style intervention in comparison to standard (control) arm. The intervention would consist of nutritional and physical activity advice.
  Consists of 5 sessions during the two years course of follow up. Three sessions in the first year (intensive phase), two sessions (maintenance phase) in second year. Overall sessions have a theme with simple selected theoretical background information. Sessions are to be interactive. Selected handouts and pamphlets are given after the session. Teaching material is both available in English and Urdu (local) language.
  Interventions: Behavioral: Life style intervention

INTERVENTIONS:
Behavioral: Life style intervention — The main goals of intervention will focus mainly on: Weight reduction ≥ 5% , moderate intensity physical activity ≥ 30 min daily, dietary fat <30 proportion of total energy, saturated fat <10%, Fiber ≥ 15g/1,000 kcal There will be 9 sessions during the two years course of follow-up
  Arms: life style intervention arm

SUMMARY:
The Karachi-based Pakistan Diabetes Prevention Study aims to address key issues in the prevention of type 2 diabetes. Approximately 20,000 people From four communities will be screened for diabetes risk factors using a non-invasive diabetes risk-score system. Those found to be at increased risk will be given an oral glucose tolerance test. People who, after the oral glucose tolerance test, are identified as having prediabetes or normal but with risk factors such as raised BMI and/or history of hypertension will have the opportunity to take part in the Pakistan Diabetes Prevention Study lifestyle intervention. This consists of culturally adjusted preventive strategies focusing on diet and physical activity in real-life settings. Another important aspect of this trial will be to assess the impact of urban planning on the prevalence of obesity and diabetes.

DETAILED DESCRIPTION:
The aim of this study is to translate the life style intervention project to prevent diabetes into real life settings in Karachi, Pakistan, home to one sixth of the world's population.

ELIGIBILITY:
Inclusion Criteria:

-Adult men and women between 30-64 years of age

Exclusion Criteria:

* Diagnosed type 1 or type 2 diabetes
* Pregnancy or presence of chronic disease rendering survival for three years unlikely
* Any psychological or physical disability to interfere with participation in the study
* Ischemic heart disease

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1564 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Type 2 Diabetes | 2 yrs
  Incidence of type 2 diabetes based on OGTT, diagnosed by WHO criteria at interim and end of an intervention.

SECONDARY OUTCOMES:
Components of Metabolic syndrome | 2 years
  To assess the difference in incidence of components of metabolic syndrom which includes waist circumference, dyslipidimia, blood pressure etc between control and intervention arm after 2 years of lifestyle intervention.
The impact of city planning on prevalence of obesity and type 2 diabetes | 2 years
  The communities will be divided according to number and accessibility of parks. The community with large number of parks will be compared with community with no parks and then change in incidence of diabetes and obesity after 2 years of lifestyle intervention will be assessed and compared between two communities. By this it would be feasible to convince local authorities to incorporate this into their agenda for future urban design.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Ahmed, MRCP(UK), Principal Investigator — The Aga Khan University Hospital; Jaweed Akhter, FRCP, Principal Investigator — The Aga Khan University Hospital
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided